CLINICAL TRIAL: NCT06268665
Title: A Randomized Trial of Tart Cherry Juice as a Dietary Supplement for the Prevention of Paclitaxel-Induced Neuropathy
Brief Title: Tart Cherry Juice as a Dietary Supplement for the Prevention of Paclitaxel-Induced Neuropathy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eve Rodler (Other)
Responsible Party: Sponsor-Investigator, Eve Rodler, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCDCC307; NCI-2024-02360 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCDCC307 (Other: University of California Davis Comprehensive Cancer Center)
Record Dates: First submitted 2024-02-02; First posted 2024-02-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer; Breast Cancer Stage I; Breast Cancer Stage II; Breast Cancer Stage III; Breast Cancer Stage IV; Invasive Breast Cancer; Ovarian Cancer; Ovarian Cancer Stage 1; Ovarian Cancer Stage II; Ovarian Cancer Stage III; Ovarian Cancer Stage IV; Ovarian Cancer Stage IA; Ovarian Cancer Stage IB; Ovarian Cancer Stage IC; Ovarian Cancer Stage 2; Ovarian Cancer Stage 3; Ovarian Cancer Stage IIIb; Ovarian Cancer Stage IIIC; Breast Cancer Stage IIIA; Breast Cancer Invasive; Breast Cancer, Stage IA; Breast Cancer, Stage IB; Breast Cancer Stage IIA; Breast Cancer Stage IIB; Breast Cancer Stage IIIB; Breast Cancer Stage IIIc; Cancer, Breast; Tumors, Breast; Mammary Cancer; Mammary Carcinoma; Breast Carcinoma; Breast Neoplasm; Malignant Breast Neoplasm; Malignant Tumor of Breast; Cancer of Ovary; Ovary Cancer; Ovary Neoplasm
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: High-Dose Tart Cherry Juice Supplement (Experimental): 1 oz tart cherry juice concentrate diluted in water up to 8oz.
  Interventions: Drug: Tart Cherry Juice
- Arm 2: Low-Dose Tart Cherry Juice Supplement (Experimental): ¼ oz tart cherry juice concentrate diluted in water up to 8oz.
  Interventions: Drug: Tart Cherry Juice

INTERVENTIONS:
Drug: Tart Cherry Juice — Given PO
  Other Names: Juice extracted from Montmorency cherries; Juice from Prunus cerasus

SUMMARY:
This is a single institution phase II randomized study evaluating the potential benefits of a supplement, tart cherry juice at high- versus low-doses, to prevent taxane induced peripheral neuropathy in breast and ovarian cancer patients undergoing paclitaxel chemotherapy.

Eligible participants enrolled onto the study will be block randomized in a 1:1 allocation to either the tart cherry juice high-dose group (Arm 1) or the tart cherry juice low-dose group (Arm 2).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE: I. Efficacy of tart cherry juice supplementation in the prevention of paclitaxel-induced peripheral neuropathy (PIPN) in breast and ovarian cancer patients undergoing treatment with paclitaxel-based chemotherapy.

SECONDARY OBJECTIVE:

I. Compare the effectiveness of high- dose and low-dose tart cherry juice supplement in reducing the severity of PIPN in breast and ovarian cancer patients undergoing treatment with paclitaxel-based chemotherapy.

II. Assess the impact of tart cherry juice on dose delivery of taxane chemotherapy.

III. Ascertain the tolerability and side effects of intake of high-dose and low-dose tart cherry juice OUTLINE: Tart cherry juice in both arms must begin ≤ 7 days from start of taxane therapy. During treatment, each participant in the high-dose group will consume 1 oz of tart cherry juice twice per day for up to 14 weeks (maximum cumulative volume of 196 oz). Each participant in the low-dose group will consume ¼ oz of tart cherry juice twice per day for up to 14 weeks (maximum cumulative volume of 49 oz). Participants will have follow-up visits at the conclusion of chemotherapy and at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive breast or ovarian cancer (Stage I, II, III, or IV) as per AJCC 8th Edition, 2018 Staging Criteria.
* Must be planning to receive paclitaxel weekly for 12 weeks (12 weeks total) as part of neoadjuvant, adjuvant, or metastatic cancer treatment.

  * Concurrent biologic therapy (e.g., trastuzumab and pertuzumab) is allowed.
  * Currently receiving hormone therapy, bisphosphonates, denosumab or LHRH-agonists is allowed.
  * Concurrent use of immune checkpoint inhibitor therapy is allowed.
  * (Neo)adjuvant chemotherapy with doxorubicin and cyclophosphamide is allowed.
  * Concurrent use of carboplatin with weekly paclitaxel in the study is allowed.
* May participate concurrently in other cancer trials.
* Must be able to complete questionnaires in English or Spanish.
* Age ≥ 18 years old at the time of consent.
* ECOG performance status of 0 - 1 (Karnofsky scale ≥ 70%, see Appendix).
* Ability to understand and the willingness to sign a written informed consent document.
* Individuals of child-bearing potential must agree to use birth control (e.g., hormonal or barrier method; abstinence, an intrauterine device) prior - to study entry, for the duration of study participation (including dose interruptions), and for 3 months after the last dose of tart cherry juice supplement; or be surgically sterilized (e.g., hysterectomy or tubal ligation).
* Patients with known human immunodeficiency virus (HIV) are allowed in the study, but HIV-positive patients must have:

  * A stable regimen of highly active anti-retroviral therapy (HAART)
  * No requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections
  * A CD4 count above 250 cells/µL and an undetectable HIV viral load on standard PCR-based tests within the last year.
* Stated willingness to not drink any additional tart cherry or any cherry juice while on the study.
* Ability and willingness to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

* Have received any prior therapy with taxanes, vinca alkaloids, eribulin, ixabepilone, or platinum. Doxorubicin is allowed (≥ 2 week washout period required).
* Active or history of peripheral neuropathy, or any chronic diseases associated with peripheral neuropathy such as diabetes mellitus, alcohol use disorder, or systemic lupus erythematosus.
* Currently taking anticoagulant medication.
* Currently taking Vitamin E, glutamine, alpha lipoic acid, gabapentin, nortriptyline, amitriptyline or duloxetine. If a patient is taking any of these supplements/medications, they must agree to stop at the time of registration. Multivitamins containing Vitamin E are allowed, however Vitamin E > 1,000 international units (IU) must be discontinued at the time of registration.
* Patients may not use cold therapy gloves for chemotherapy induced neuropathy.
* Known allergy to cherries.
* Inability to swallow liquid.
* Pregnant or breastfeeding individuals (lactating individuals must agree not to breast feed while taking study juice supplementation).
* Any condition that would prohibit the understanding or rendering of informed consent.
* Any condition that in the opinion of the investigator would interfere with safety or compliance while on trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of tart cherry juice supplementation in the prevention of paclitaxel-induced peripheral neuropathy (PIPN) in breast and ovarian cancer patients undergoing treatment with paclitaxel-based chemotherapy. | Up to 1 year.
  Number of participants between study arms experiencing PIPN using the 11-item peripheral neuropathy component of the Functional Assessment of Cancer Therapy-Taxane (FACT-Taxane) survey.

SECONDARY OUTCOMES:
Compare the effectiveness of high- dose and low-dose tart cherry juice supplement in reducing the severity of PIPN in breast and ovarian cancer patients undergoing treatment with paclitaxel-based chemotherapy. | Up to 1 year.
  Assessment of the severity of PIPN using the Functional Assessment of Cancer Therapy-Taxane (FACT-Taxane) neuropathy subscale survey and National Cancer Institute Common Terminology Criteria for Adverse Events version 5 (NCI CTCAE v.5) physician assessment.
Assess the impact of tart cherry juice on dose delivery of taxane chemotherapy. | Up to 1 year.
  Number of participants between arms experiencing dose reductions, delays, or discontinuations.
Tolerability of daily intake of high-dose and low-dose tart cherry juice. | Up to 1 year.
  Number of participants between study arms ≥90% compliant with daily consumption of tart cherry juice.
Safety profile of daily intake of high-dose and low-dose tart cherry juice. | Up to 1 year.
  Number of participants between study arms with adverse events graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE v5).

CONTACTS AND LOCATIONS:
Overall Officials: Eve Rodler, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States